CLINICAL TRIAL: NCT03790371
Title: Vaginal Misoprostol Before Intrauterine Contraceptive Device Insertion Following Previous Insertion Failure
Brief Title: Vaginal Misoprostol Before Intrauterine Contraceptive Device Insertion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ain Shams University MH
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Contraception
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- misoprostol group (Active Comparator): misoprostol (misotac® sigma pharmaceutical industries) 200 mcg vaginally applied ten and four hours prior to the second attempt of IUD insertion
  Interventions: Drug: Misoprostol
- placebo (Placebo Comparator): while the control group received a placebo tablet in the same regimen as the study group.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Misoprostol — vaginal misoprostol prior IUD insertion
  Arms: misoprostol group
Drug: Placebos — vaginal placebo tablet prior IUD insertion
  Arms: placebo

SUMMARY:
the current study was conducted to assess efficacy of vaginal misoprostol before IUD insertion following previous insertion failure

ELIGIBILITY:
Inclusion Criteria:

One previous failed attempt of IUD insertion.

Exclusion Criteria:

1. Uterine fibroid distorting the cavity.
2. Anatomical uterine abnormality with distortion of the cavity
3. Current pelvic inflammatory disease or recently treated pelvic inflammatory disease (PID) in the last three months.
4. Current purulent cervicitis (chlamydia or gonorrhea).
5. Immediately after septic abortion.
6. Uterus size less than 6 cm and more than 9 cm.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
the success rate for IUD insertion. | four hours after misoprostol dose
  the success of IUD insertion after previous attempt failure

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt